CLINICAL TRIAL: NCT02146339
Title: Impact of Milk Polar Lipids Content in a Test Meal on Lipid Composition of Ileostomy Fluid and Consequences on Postprandial Dietary Cholesterol and Fatty Acid Metabolism.
Brief Title: Impact of Milk Polar Lipids on Lipids Digestion, Absorption and Metabolism
Acronym: VALOBAB-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013.828
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cardiometabolic Risk
Keywords: nutrition; milk; polar lipids; cardiometabolic risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Unfortified-3g-5g milk polar lipid fortified cheese product (Experimental): Each subject will receive a single dose of each cheese product (100 g) containing no or 3g or 5g of milk polar lipids, 300 mg of [1,1,1]-13C-triolein and 45 mg of 2H6-cholesterol. The wash-out period is four weeks.
  Interventions: Other: Cheese n°1- cheese n°2 - cheese n°3
- Unfortified-5g-3g milk polar lipid fortified cheese product (Experimental): Each subject will receive a single dose of each cheese product (100 g) containing no or 3g or 5g of milk polar lipids, 300 mg of [1,1,1]-13C-triolein and 45 mg of 2H6-cholesterol. The wash-out period is four weeks.
  Interventions: Other: Cheese n°1- cheese n°3 - cheese n°2
- 3g-5g milk polar lipid fortified-unfortified cheese product (Experimental): Each subject will receive a single dose of each cheese product (100 g) containing no or 3g or 5g of milk polar lipids, 300 mg of [1,1,1]-13C-triolein and 45 mg of 2H6-cholesterol. The wash-out period is four weeks.
  Interventions: Other: Cheese n°2- cheese n°3 - cheese n°1
- 3g-Unfortified-5g milk polar lipid fortified cheese product (Other): Each subject will receive a single dose of cheese n°1, then cheese n°2 after a wash-out period of 4 weeks, then cheese n°3 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Interventions: Other: cheese n°2 - cheese n°1- cheese n°3
- 5g-unfortified-3g milk polar lipid fortified cheese product (Experimental): Each subject will receive a single dose of each cheese product (100 g) containing no or 3g or 5g of milk polar lipids, 300 mg of [1,1,1]-13C-triolein and 45 mg of 2H6-cholesterol. The wash-out period is four weeks.
  Interventions: Other: Cheese n°3 - cheese n°1- cheese n°2
- 5g-3g milk polar lipid fortified-unfortified cheese product (Other): Each subject will receive a single dose of each cheese product (100 g) containing no or 3g or 5g of milk polar lipids, 300 mg of [1,1,1]-13C-triolein and 45 mg of 2H6-cholesterol. The wash-out period is four weeks.
  Interventions: Other: Cheese n°3- cheese n°2 - cheese n°1

INTERVENTIONS:
Other: Cheese n°1- cheese n°2 - cheese n°3 — Each subject will receive a single dose of cheese n°1, then cheese n°2 after a wash-out period of 4 weeks, then cheese n°3 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: Unfortified-3g-5g milk polar lipid fortified cheese product
Other: Cheese n°1- cheese n°3 - cheese n°2 — Each subject will receive a single dose of cheese n°1, then cheese n°3 after a wash-out period of 4 weeks, then cheese n°2 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: Unfortified-5g-3g milk polar lipid fortified cheese product
Other: cheese n°2 - cheese n°1- cheese n°3 — Each subject will receive a single dose of cheese n°2, then cheese n°1 after a wash-out period of 4 weeks, then cheese n°3 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: 3g-Unfortified-5g milk polar lipid fortified cheese product
Other: Cheese n°2- cheese n°3 - cheese n°1 — Each subject will receive a single dose of cheese n°2, then cheese n°3 after a wash-out period of 4 weeks, then cheese n°1 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: 3g-5g milk polar lipid fortified-unfortified cheese product
Other: Cheese n°3 - cheese n°1- cheese n°2 — Each subject will receive a single dose of cheese n°3, then cheese n°1 after a wash-out period of 4 weeks, then cheese n°2 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: 5g-unfortified-3g milk polar lipid fortified cheese product
Other: Cheese n°3- cheese n°2 - cheese n°1 — Each subject will receive a single dose of cheese n°3, then cheese n°2 after a wash-out period of 4 weeks, then cheese n°1 after a wash-out period of 4 weeks.
  Cheese n°1 = unfortified cheese product Cheese n°2 = 3 g milk polar lipid fortified cheese product Cheese n°3 = 5 g milk polar lipid fortified cheese product
  Arms: 5g-3g milk polar lipid fortified-unfortified cheese product

SUMMARY:
Polar lipids have a specific chemical structure: they are an essential component of human cell membranes, play a major role in the nervous system and also influence the metabolic pathways including the cholesterol metabolism.

Polar lipids are used in food-processing industry for their emulsification properties. The most famous emulsifier is soya lecithin but milk also naturally contains natural emulsifiers such as polar lipids. Milk polar lipids are rich in sphingomyelin and they may have beneficial effects on lipid metabolism in the context of metabolic diseases of nutritional origin.

The purpose of this research is to study the variation of sphingomyelin content at the ileum's end after the consumption of different doses of milk polar lipids, and consequences on the intestinal absorption and metabolism of fatty acids and cholesterol.

The subjects will be taking three different test meals varying by their milk polar lipids content.

It is a bi-centric study with a centre in LYON (Centre de Recherche en Nutrition Humaine Rhône-Alpes) and CLERMONT-FERRAND (Centre de Recherche en Nutrition Humaine Auvergne).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 75 years
* Having undergone a temporary or permanent ileostomy,
* Considered to have well-functioning ileostomy
* Normal (or not clinically significant) lipid parameters

Exclusion Criteria:

* Ileostomy due to an ongoing digestive cancer
* Ileostomy due to a Chrohn's disease
* Dairy products allergy or intolerance
* Medication that could interfere with lipid metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Ileal sphingomyelin output | up to Day 63
  The total sphingomyelin output will be measured in the ileostomy fluids over 8 hours after the consumption of the 3 different test meals.

SECONDARY OUTCOMES:
Plasma lipids and isotopic tracers | A least Day 7, Day 35 and Day 63
  Plasma lipids and isotopic tracers will be measured after the consumption of the 3 different test meals. Fasting and postprandial measurements over 8 hours depending on parameters.
Plasma glucose and insulin | At least Day 7, Day 35 and Day 63
  Plasma glucose and insulin will be measured after the consumption of the 3 different test meals. Fasting and postprandial measurements over 8 hours.
Energy expenditure and substrate oxidation with indirect calorimetry | At least Day7, Day 35 and Day 63
  Energy metabolism and 13CO2 will be measured after the consumption of the 3 different test meals. Fasting and during all the postprandial period (8 h).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de recherche en Nutrition Humaine-Auvergne -Unité d'Exploration Nutritionnelle, Clermont-Ferrand
  - Centre de Recherche en Nutrition Humaine Rhône-Alpes, Lyon

REFERENCES:
- [Derived] Le Barz M, Vors C, Combe E, Joumard-Cubizolles L, Lecomte M, Joffre F, Trauchessec M, Pesenti S, Loizon E, Breyton AE, Meugnier E, Bertrand K, Drai J, Robert C, Durand A, Cuerq C, Gaborit P, Leconte N, Bernalier-Donadille A, Cotte E, Laville M, Lambert-Porcheron S, Ouchchane L, Vidal H, Malpuech-Brugere C, Cheillan D, Michalski MC. Milk polar lipids favorably alter circulating and intestinal ceramide and sphingomyelin species in postmenopausal women. JCI Insight. 2021 May 24;6(10):e146161. doi: 10.1172/jci.insight.146161. PMID 33857018
- [Derived] Vors C, Joumard-Cubizolles L, Lecomte M, Combe E, Ouchchane L, Drai J, Raynal K, Joffre F, Meiller L, Le Barz M, Gaborit P, Caille A, Sothier M, Domingues-Faria C, Blot A, Wauquier A, Blond E, Sauvinet V, Gesan-Guiziou G, Bodin JP, Moulin P, Cheillan D, Vidal H, Morio B, Cotte E, Morel-Laporte F, Laville M, Bernalier-Donadille A, Lambert-Porcheron S, Malpuech-Brugere C, Michalski MC. Milk polar lipids reduce lipid cardiovascular risk factors in overweight postmenopausal women: towards a gut sphingomyelin-cholesterol interplay. Gut. 2020 Mar;69(3):487-501. doi: 10.1136/gutjnl-2018-318155. Epub 2019 Jun 12. PMID 31189655
- See also: Related Info — http://www.crnh-rhone-alpes.fr
- See also: Related Info — http://www1.clermont.inra.fr/crnh/